## Assessment of Quality of Life Changes on Lower Extremity Lymphedema Patients using an Advanced Pneumatic Compression Device at Home.

Protocol# 5010

03 July 2019 Protocol Version 3.1

# **Investigator Signature**

| Protocol Title: Assessment of Quality of Life<br>Patients using a Pneumatic Compression Dev | |
|---|---|
| Protocol Number: 5010 | |
| Date: 03 July 2019, Version 3.1 | |
| I confirm that I have read this protocol. I will Good Clinical Practices (GCP), institutional rappropriate regulatory requirements. | l comply with the protocol and the principles of research policies and procedures and other |
| Site Principal Investigator Name (Print) | |
| Site Principal Investigator Signature | Date |

## **SYNOPSIS**

| Title of Study | Assessment of Quality of Life Changes on Lower Extremity Lymphedema Patients |
|---|---|
| | using an Advanced Pneumatic Compression Device at Home. |
| Protocol Date | 3 July 2019 |
| Protocol Version | 3.1 |
| Name of Sponsor | Tactile Medical™ |
| Device | Flexitouch® system or Flexitouch® Plus |
| Primary Endpoint | Quality of life (QoL), lymphedema symptoms, lymphedema and venous related complication rate, lymphedema and venous related unscheduled visits |
| Secondary Endpoint | Limb circumference changes, Flexitouch compliance, skin changes, QoL |
| METHODOLOGY | |
| Study Design | Multi-center, single arm, observational clinical trial |
| Treatments | Subjects will be instructed to use the Flexitouch system or Flexitouch Plus as prescribed and will be followed for 52 weeks. The subjects will be seen in clinic 4, 8, 12, 24 and 52 weeks after completion of device training. The subject will also have phone call follow-ups at 1, 18, 32 and 40 weeks after device training. |
| <b>Treatment Duration</b> | As prescribed |
| SUBJECT POPULATION | |
| Number Planned | 300 |
| Inclusion Criteria | <ol> <li>Age 18 or older</li> <li>Diagnosis of primary or secondary, unilateral or bilateral, LE lymphedema</li> <li>Ability and willingness to participate in all aspects of the study including following prescribed care</li> <li>Ability to provide informed consent</li> <li>Must have a prescription for the Flexitouch (Flexitouch system or Flexitouch Plus)</li> </ol> |
| Exclusion Criteria | <ol> <li>Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy or primary surgery for the treatment of cancer.</li> <li>Active skin or limb infection/inflammatory disease (acute cellulitis, or other uncontrolled skin or untreated inflammatory skin disease)</li> <li>Acute thrombophlebitis (in last 2 months)</li> <li>Pulmonary embolism within the previous 6 months</li> <li>Deep Vein Thrombosis (DVT) within the previous 3 months</li> <li>Severe peripheral artery disease (critical limb ischemia including ischemic rest pain, arterial wounds, or gangrene)</li> <li>Pulmonary edema</li> <li>Heart failure (acute pulmonary edema, decompensated acute heart failure)</li> <li>Patients with poorly controlled asthma</li> <li>Previous use of the study pneumatic compression device (PCD)</li> <li>Currently using multi-layer bandaging (MLB) unless bandages can be removed for limb circumference measurements</li> <li>Pregnant women or women of childbearing potential not on contraception</li> <li>Any condition where increased venous and lymphatic return is undesirable</li> <li>Currently participating in another medical device or drug clinical trial</li> <li>Signs of noncompliance at the week 4 visit, including: using the device less than 3 times per week and/or not attending the scheduled visit</li> </ol> |

#### **Table of Contents**

| Invest | igator s | Signature | 2 |
|---|---|---|---|
| SYNOI | PSIS | | 3 |
| 1.0 | Conta | ct Information | 7 |
| 1.1 | Spo | onsor Contact Information | 7 |
| 1.2 | Stu | dy Principal Investigator Information | 7 |
| 2.0 | Abbre | eviations | 7 |
| 3.0 | Intro | luction | 7 |
| 3.1 | Bad | kground and Rationale | 7 |
| 3.2 | De | vice Description | 8 |
| 4.0 | Study | Objectives | 8 |
| 5.0 | Study | Design | 8 |
| 5.1 | Stu | dy Endpoints | 9 |
| 5 | .1.1 | Primary Endpoints | 9 |
| 5 | .1.2 | Secondary Endpoints | 9 |
| 5.2 | Suk | eject Selection | 10 |
| 5 | .2.1 | Inclusion Criteria | 10 |
| 5 | .2.2 | Exclusion Criteria | 10 |
| 5 | .2.3 | Subject Withdrawal or Early Termination | 11 |
| 5.3 | Do | sage and Rationale | 11 |
| 5.4 | Stu | dy Timetable | 11 |
| 6.0 | Study | Visit Summaries | 11 |
| 6.1 | Scr | eening/Baseline Visit | 11 |
| 6.2 | We | ek 0/Training | 12 |
| 6.3 | We | eks 1 (+7 days), 18, 32, & 40 (± 14 days) Follow-up Phone Calls | 12 |
| 6.4 | We | eks 4, 8, 12 (± 7 days), 24, and 52 (± 14 days) In-Clinic Follow-Up Visit(s) | 12 |
| 7.0 | Study | Procedures | 12 |
| 7.1 | Info | ormed Consent | 12 |
| 7.2 | De | mographics & Medical History | 13 |
| 7.3 | Vit | al Signs | 13 |
| 7.4 | Ski | n Assessment | 13 |

| 7. | .4.1 | Fibrosis Grading | 13 |
|---|---|---|---|
| 7. | .4.2 | Assessment of Skin Changes | 13 |
| 7. | .4.3 | Lymphedema Staging | 14 |
| 7.5 | Lim | b Circumference Measurements | 14 |
| 7. | .5.1 | Mark Anatomical Sites | 14 |
| 7. | .5.2 | Circumference Measurements | 15 |
| 7.6 | Pho | otograph (Legs) | 15 |
| 7.7 | Pre | scribed Care & Treatment Protocol | 16 |
| 7.8 | Me | dication Review | 16 |
| 7.9 | Qol | L Questionnaires | 16 |
| 7.10 | ) Flex | kitouch Compliance Assessment & Subject Diary | 17 |
| 7.11<br>Obs | | nphedema and Venous Related HCU, Device-Related Adverse Events, & Device | 17 |
| 7. | .11.1 | Lymphedema and Venous Related HCU | 17 |
| 7. | .11.2 | Device-Related Adverse Events | 18 |
| 7. | .11.3 | Device Observations | 18 |
| 7.12 | . Flex | xitouch Administration & Training | 18 |
| 7.13 | Stu | dy Schedule of Activities | 19 |
| 8.0 | Study | Device Accountability | 20 |
| 9.0 | Risk A | nalysis and Adverse Events | 20 |
| 9.1 | Risk | < Analysis | 20 |
| 9.2 | Adv | verse Events | 20 |
| 10.0 | Deviat | tion from Study Plan | 20 |
| 11.0 | Qualit | ry Assurance Procedures | 20 |
| 11.1 | Site | Qualification | 21 |
| 11.2 | 2 Dat | a Collection Procedures | 21 |
| 11.3 | S Clin | ical Site Monitoring | 21 |
| 11.4 | Dat | a Safety Monitoring | 21 |
| 12.0 | Chang | ge to Investigational Plan | 23 |
| 13.0 | Statist | tical Methods and Determination of Sample Size | 23 |
| 13.1 | Stat | tistical Analysis Plan | 23 |
| 13.2 | 2 Det | ermination of Sample Size | 23 |
| 14.0 | Comp | ensation | 23 |

| 15.0 | Publication Plan | 23 |
|-------|---------------------------------------------------|----|
| 16.0 | References | 23 |
| 17.0 | Appendices | 24 |
| Appei | endix A: Lymphedema Quality of Life Tool (LYMQOL) | 25 |
| Appei | endix B: SF-36 Health Survey v.2 (SF-36) | 28 |
| Appei | endix C: Subject Diary | 35 |

#### 1.0 Contact Information

## 1.1 Sponsor Contact Information

Tactile Medical<sup>TM</sup>
Jill Christensen, Clinical Research Manager
1331 Tyler Street NE, Suite 200
Minneapolis, MN 55413
612-355-5123
jchristensen@tactilemedical.com

## 1.2 Study Principal Investigator Information

Thomas Maldonado, MD New York Vascular Surgery Associates 530 First Avenue Suite F New York City, NY 10016 212.263.7311 Thomas.maldonado@nyumc.org

#### 2.0 Abbreviations

| CFR | Code of Federal Regulations |
|-------|------------------------------|
| CRA | Clinical Research Associate |
| CRF | Case Report Form |
| DVT | Deep Vein Thrombosis |
| ER | Emergency Room |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HCU | Health Care Utilization |
| IC | Informed Consent |
| IRB | Institutional Review Board |
| LE | Lower Extremity |
| MLB | Multi-Layer Bandaging |
| PCD | Pneumatic Compression Device |
| QoL | Quality of Life |
| SAE | Serious Adverse Event |
| SF-36 | Short Form-36 |

#### 3.0 Introduction

#### 3.1 Background and Rationale

The purpose of this study is to evaluate the effect of an advanced pneumatic compression device in improving symptoms and quality of life in patients with lower extremity lymphedema.

Lymphedema is a chronic and disfiguring disease usually secondary to excessive fluid and protein accumulation in the interstitium as result of lymphatic system obstruction.<sup>1</sup> It can occur either primarily (as a result of congenital malformations)

or secondarily (as a result of trauma to the lymphatic system, surgery, radiation therapy, obesity and chronic venous insufficiency).<sup>2,3</sup> This leads to limb swelling in early stages with progression to thickening skin and fibrosis leaving the affected extremity susceptible to skin breakdown and repeated infections. There is no cure for lymphedema, and the available treatment modalities consist of manual lymphatic drainage, compression therapy, and in very severe cases lymphatic exchange, a costly and invasive procedure.<sup>4</sup>

Pneumatic Compression Devices (PCDs) offer a novel modality for treatment of lymphatic obstruction. The Flexitouch® System and Flexitouch® Plus are PCDs that target all major lymphatic beds and release pressure in a systematic manner, mimicking a functional drainage system.<sup>5</sup> Prior studies demonstrated improvement in control of edema and ease of use; however improvement in quality of life (QoL) and decrease in symptoms has not been thoroughly evaluated.<sup>6,7,8</sup> Therefore we propose to demonstrate improved QoL and symptoms in patients with lower extremity (LE) lymphedema.

#### 3.2 Device Description

The Flexitouch system and Flexitouch Plus (Tactile Medical<sup>TM</sup>, Minneapolis, MN, USA) are segmental, programmable, gradient PCDs which have been cleared by the Food and Drug Administration (FDA) for market in the US (K013061), (US HCPCS code E0652). The devices consist of a controller and garment set. The garments are constructed of nylon and have 27-32 chambers, depending upon garment size. The pressure setting is variable between "normal" and "increased." The Flexitouch system and Flexitouch Plus are intended for the treatment of lymphedema, primary lymphedema, post mastectomy edema, edema following trauma and sports injuries, post immobilization edema, venous insufficiencies, reducing wound healing time and assistance in healing stasis dermatitis, venous stasis ulcers, or arterial and diabetic leg ulcers.

The Flexitouch Plus is functionally equivalent to the Flexitouch system, however it permits bilateral treatment of the lower extremities, incorporates a color display with larger buttons on the controller, and provides more comfortable garments that are easier to put on and take off.

### 4.0 Study Objectives

The study will assess QoL, lymphedema symptoms, lymphedema and venous related complication rate, lymphedema and venous related unscheduled visits, Flexitouch compliance, and skin and limb circumference changes in primary or secondary, unilateral or bilateral, lower extremity lymphedema patients using the Flexitouch system or Flexitouch Plus during the 52 week study period.

## 5.0 Study Design

This investigation is a post-market, on label, multi-center, single arm, observational clinical trial of a prospective cohort of 300 subjects with primary or secondary, unilateral or bilateral, lower extremity lymphedema in the United States. All subjects will receive PCD treatment for 52 weeks (*Figure 1*).



Figure 1. Study Design

## 5.1 Study Endpoints

#### 5.1.1 Primary Endpoints

The following primary endpoints for this study will compare changes after 12 weeks of treatment to baseline for the following parameters:

- QoL
- Lymphedema symptoms

In addition, the number of occurrences after 52 weeks of treatment will be compared to the number of occurrences in the year preceding treatment for the following variable:

• Lymphedema and venous related health care utilization

#### 5.1.2 Secondary Endpoints

The secondary endpoints for this study will compare changes after 12 and 52 weeks of treatment to baseline for the following:

- Limb circumference
- Skin evaluation

In addition, changes after 24 and 52 weeks of treatment to baseline for the following parameter:

#### QoL

To assess Flexitouch compliance, subjects will be categorized as noncompliant, partially compliant, or compliant (Table 1). Primary and secondary outcomes will then be compared across the defined compliance categories.

Table 1. Compliance Category Definitions

| <b>Compliance Category</b> | Definition |
|---|---|
| Noncompliant | Prescribed care followed an average of 0-2 days per week. |
| Partially Compliance | Prescribed care followed an average of 3-4 days per week. |
| Compliant | Prescribed care followed an average of 5-7 days per week. |

## 5.2 Subject Selection

#### 5.2.1 Inclusion Criteria

- 1. Age 18 or older
- 2. Diagnosis of primary or secondary, unilateral or bilateral, LE lymphedema
- 3. Ability and willingness to participate in all aspects of the study including following prescribed care
- 4. Ability to provide informed consent
- 5. Must have a prescription for the Flexitouch (Flexitouch system or Flexitouch Plus)

#### 5.2.2 Exclusion Criteria

- 1. Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy or primary surgery for the treatment of cancer.
- 2. Active skin or limb infection/inflammatory disease (acute cellulitis, or other uncontrolled skin or untreated inflammatory skin disease)
- 3. Acute thrombophlebitis (in last 2 months)
- 4. Pulmonary embolism within the previous 6 months
- 5. Deep Vein Thrombosis (DVT) within the previous 3 months
- 6. Severe peripheral artery disease (critical limb ischemia including ischemic rest pain, arterial wounds, or gangrene)
- 7. Pulmonary edema
- 8. Heart failure (acute pulmonary edema, decompensated acute heart failure)
- 9. Patients with poorly controlled asthma
- 10. Previous use of the study PCD

- 11. Currently using multi-layer bandaging (MLB) unless bandages can be removed for limb circumference measurements
- 12. Pregnant women or women of childbearing potential not on contraception
- 13. Any condition where increased venous and lymphatic return is undesirable
- 14. Currently participating in another medical device or drug clinical trial
- 15. Signs of noncompliance at the week 4 visit, including: using the device less than 3 times per week and/or not attending the scheduled visit

### 5.2.3 Subject Withdrawal or Early Termination

Subjects will exit the study if they meet any of the following criteria:

- Subject death
- Subject voluntarily withdraws
- Subject acquires one or more of the exclusion criteria whereby the investigator deems study discontinuation a necessity
  - If subject acquires an infection, they may be treated for the infection and continue in the trial at the investigator's discretion.
     Detailed information regarding the infection, nature, treatment, and duration will be recorded.
- Subject diary shows an unwillingness to remain partially compliant or compliant with prescribed care (subject will be considered a screen failure if he or she uses the device <3 times per week on average at the Week 4 visit).

## 5.3 Dosage and Rationale

Study subjects will be instructed to conduct LE treatment as prescribed by their physician. They will also be instructed to wear clinically appropriate compression garments and participate in proper skin care as part of their routine care.

#### 5.4 Study Timetable

Table 2. Study Timetable

| | 1-6 months | 7-12 months | 12-24 months | 24-36 months |
|------------------|------------|-------------|--------------|--------------|
| IRB Review | X | | | |
| Enrollment | X | X | X | X |
| Treatment | X | X | X | X |
| Data Entry | X | X | X | X |
| Data Analysis | | | | X |
| Manuscript Draft | | | | X |
| Publication | | | | 2021 |

#### **6.0** Study Visit Summaries

The sections below provide a summary of procedures at each study visit. For further detail for each procedure, please refer to section 7 (Study Procedures) of the protocol.

In the event a patient is unwilling or unable to attend a scheduled Follow-Up Visit, the site will have the discretion to offer a home visit to the patient.

### 6.1 Screening/Baseline Visit

Informed Consent Discussion

- Inclusion/Exclusion criteria assessment
- Collection of demographics, significant medical history, and lymphedema history
- Urine pregnancy test (as applicable)
- Weight (kg) and height (cm)
- Skin assessment
- Limb circumference
- Photographs (Leg)
- Prescribed care and treatment protocol
- Medication review
- Qol Questionnaires
  - o SF-36
  - o LYMQOL
- Subject Diary (dispense)

## 6.2 Week 0/Training

• The subject will receive the Flexitouch system or Flexitouch Plus and be instructed on use from a Tactile Medical trainer. Device treatment will commence following the visit from the trainer.

#### 6.3 Weeks 1 (+7 days), 18, 32, & 40 (± 14 days) Follow-up Phone Calls

- Prescribed care and treatment protocol
- Medication review
- Flexitouch compliance assessment
- Complication, adverse event, and device observation assessment

## 6.4 Weeks 4, 8, 12 (± 7 days), 24, and 52 (± 14 days) In-Clinic Follow-Up Visit(s)

- Weight (kg)
- Skin assessment
- Limb circumference
- Photographs (Leg)
- Prescribed care and treatment protocol
- Medication review
- QoL Questionnaires (Weeks 12, 24, and 52 only)
  - o LYMOOL
  - o SF-36
- Subject diary collection
- Flexitouch compliance assessment
- Complication, adverse event, and device observation assessment

#### 7.0 Study Procedures

#### 7.1 Informed Consent

Signed consent for participation in this study will be obtained prior to any research procedures. All study participants are required to sign an Intuitional Review Board

(IRB) approved informed consent document that outlines the purpose of the study, requirements for participation, risks and benefits to participation, and subject's rights. Adequate time will be given for patients to read the consent form, to confirm their comprehension, and to decide on consent. Comprehension and capacity for consent will be assessed by the research staff.

The study staff will ensure that a valid consent is documented and placed in the patient's medical chart. A signed copy will be given to the subject/authorized representative and a copy will be maintained in the study file.

## 7.2 Demographics & Medical History

Demographics will be collected at baseline including the date of birth, ethnicity, race, gender, and employment status.

If the subject is female and of childbearing potential, a urine pregnancy test will be performed to ensure the subject is not pregnant. Per exclusion criterion 11, if a subject is pregnant or a women of childbearing potential not on contraception, they will be excluded from the study.

Significant medical history and lymphedema history will be collected at baseline including number of lymphedema and venous related visits that required health care utilization (HCU) (includes clinic visits, hospitalization, walk-in clinic/urgent care, and ER visits).

### 7.3 Vital Signs

At the screening/baseline visit, height (cm) and weight (kg) will be collected. Weight will be collected at all other clinic visit follow-ups.

#### 7.4 Skin Assessment

Skin will be assessed at each clinic visit by fibrosis grading, assessment of skin changes, and staging of lymphedema using ISL guidelines.

## 7.4.1 Fibrosis Grading

Fibrosis grading will use the following guidelines:

- Grade 0: Latent with no evident fibrosis
- <u>Grade 1</u>: Soft tissues responds only minimally or moderately to elevation (raising the limb) or compression; texture is moderately firm or spongy
- <u>Grade 2</u>: Marked increase in density and firmness; "tethering" of skin (changes in texture that makes skin look as it is being pulled from within)
- Grade 3: Very marked density and firmness with evident tethering

#### 7.4.2 Assessment of Skin Changes

The assessment of skin changes will be done by recording the presence or absence of:

- Hyperpigmentation, Discoloration
- Hyperkeratosis

- Dermatitis, Eczema
- Ulceration, Blisters
- Positive Stemmer Sign
- Squaring of Toes
- Deep Creasing at Flexion Points
- Papillomas
- Puffy Forefoot/Swelling on Dorsum
- Increase of Fat or Muscle Bulk
- Lymphorrhea, Weeping Edema

### 7.4.3 Lymphedema Staging

The staging of lymphedema will follow ISL guidelines as shown in Table 3.

Table 3. ISL Staging Guidelines

| Stage | Description |
|---|---|
| Stage 0 | Latent with no clinical signs (no evident swelling). |
| Stage 1 | Soft swelling (pitting) that resolves with elevation. |
| Stage 2 | Spongy swelling (pitting and non-pitting) that does not resolve with elevation; fibrosis may or may not be present. |
| Stage 3 | Symptoms of lymphostatic elephantitis where pitting is absent and tropic skin changes develop; extensive fibrotic swelling, blistering, ulceration, lymphorrea, papilloma, and/or recurrent infections may be present. |

## 7.5 Limb Circumference Measurements

Limb circumference measures will be taken at each in-clinic visit for both legs. The circumference measurements will be completed by research personnel with documented training showing the individual was able to independently and accurately conduct the measurements. Measurements will be collected using a Gulick II tape measure provided by Tactile Medical. In addition, if possible, the same clinician will be asked to take the measurements for each subject serially.

Standard limb measurement will involve taking two circumference measurements at 18 cm from the floor and 10 cm above the popliteal.

#### 7.5.1 Mark Anatomical Sites

Using a pen or skin marker, with the subject standing upright and bearing weight on the limb being measured, mark the subject at the lateral aspect of the leg 18 cm from the floor (see Figure 2), at the popliteal, and 10 cm from the popliteal (Figure 3).



Figure 2. Site A is 18 cm from the floor on lateral aspect of the leg.



Figure 3. Site B is the popliteal and Site C is 10 cm above the popliteal.

#### 7.5.2 Circumference Measurements

After marking the anatomical sites, measure and record the circumference, in cm, at sites A (see Figure 4) and C (see Figure 5). The tape measure must be placed precisely over (covering) the skin marking. Adjust the tension of the tape measure so that one red ball is visible in the tension indicator and record the circumference measurement.



Figure 4. Site A circumference measurement.



Figure 5. Site C circumference measurement.

### 7.6 Photograph (Legs)

A digital photograph of the subject's legs will be taken at each study visit. The subject's legs should be exposed, at minimum, from the bottom of the ankle to the mid-thigh. Subjects should sit and straighten their legs as much as possible (see Figure 6).



Figure 6. Leg photograph example.

Additionally, if a subject has areas of hyperpigmentation, ulcers, or excessive swelling, a close-up photo of that area should be taken. The image number(s) from the digital camera should be recorded on the subject's source documentation.

#### 7.7 Prescribed Care & Treatment Protocol

At each visit, current lymphedema treatment, including Flexitouch treatment, will be reviewed and recorded.

#### 7.8 Medication Review

At each clinic visit, use of the following medications will be documented:

- Beta blockers
- Diuretics
- Oral steroids
- Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)

#### 7.9 QoL Questionnaires

The LYMQOL is an assessment tool designed for measuring QoL in patients with lower limb lymphedema. It is a 25 item questionnaire which has been designed and validated in patients with chronic edema and covers 4 domains: function, appearance, symptoms, and mood and in addition has an overall QoL score. This tool has been designed and validated for patients with chronic lymphedema in one or both legs to measure QoL. (Appendix A)

The Short Form-36 (SF-36) is an assessment of functional status and quality of life. The SF-36 is a validated QoL tool that has been widely utilized and has been found to be appropriate for use in evaluating health related quality of life impacts. The SF-36 consists of 36 questions that evaluate eight health concepts including physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning – emotional, and mental health. (Appendix B)

### 7.10 Flexitouch Compliance Assessment & Subject Diary

At each phone call and clinic visit, subject compliance will be assessed by collecting the following information:

- Days Flexitouch used in past week
- Days compression garments used in past week
- Difficulty in following treatment
- Difficulty in putting on Flexitouch garments
- Difficulty using Flexitouch controller
- Pain or discomfort experienced when using Flexitouch
- Position treatment being done in

If the subject reports difficulty following treatment, putting on the Flexitouch garment, difficulty using the Flexitouch controller, or is experiencing pain or discomfort when using Flexitouch, the site may refer the subject to Tactile Medical clinical services for assistance in addressing the issue(s).

In addition, the subjects will be provided with a Subject Diary at their Screening/Baseline visit and be instructed to begin completing the diary when they start using their device after their training visit. The subject will be asked to keep a daily record of their use of Flexitouch, Actitouch (if prescribed), and compression stockings. (Appendix C) Subjects should bring their diary into each study visit for review and collection.

If the subject is noncompliant or partially compliant in device use, (see Table 1), the site should identify barriers to compliance and determine if additional device training by the site or Tactile personnel is warranted. If noncompliance continues, the Investigator may initiate the subject's withdrawal from the study.

At the 4 week in-clinic follow-up visit, if a subject is not using their Flexitouch an average of 3 times per week, they will be considered a screen failure.

If the subject experiences a complication (e.g., active infection, DVT) that requires temporary discontinuation of device use and 4 weeks of continuous treatment is not possible before the final in-clinic visit takes place, the subject should be withdrawn from the study.

Additionally, a device history log may be downloaded periodically from Flexitouch Plus units.

# 7.11 Lymphedema and Venous Related HCU, Device-Related Adverse Events, & Device Observations

At each phone call and clinic follow-up visit, assessment of lymphedema and venous related HCU, device-related adverse events, and device observations will occur and be recorded in Clindex, per the following definitions.

#### 7.11.1 Lymphedema and Venous Related HCU

Lymphedema and venous related visits that required HCU (includes clinic visits, hospitalization, walk-in clinic/urgent care, and ER visits).

#### 7.11.2 Device-Related Adverse Events

Any untoward medical occurrence in a subject that is associated with the use of the Flexitouch device.

#### 7.11.3 Device Observations

All subject-reported user errors, device failures, malfunctions, or device issues.

## 7.12 Flexitouch Administration & Training

After the subject's screening/baseline visit, Tactile Medical personnel will perform in-home device training. The date of device training (Day 0) will be used to determine the timing of subsequent follow-up visits.

## 7.13 Study Schedule of Activities

| Assessments | Screening/Baseline | Training / Day 0 | Week 1 (Phone Call) | Week 4 | Week 8 | Week 12 | Week 18 (Phone call) | Week 24 | Week 32 (Phone call) | Week 40 (Phone call) | Week 52 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window | N/A | N/A | +7 <b>Days</b> | ±7 Days | ±7 days | ±7 days | ±14 days | ±14days | ±14 days | ±14 days | ±14 days |
| Informed Consent | X | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical History/Status | $X^1$ | | | | | | | | | | |
| Vital Signs <sup>2</sup> (Height, Weight) | X | | | X | X | X | | X | | | X |
| Skin Assessment | X | | | X | X | X | | X | | | X |
| Limb Circumference | X | | | X | X | X | | X | | | X |
| Photograph (Leg) | X | | | X | X | X | | X | | | X |
| Prescribed Care & Treatment<br>Protocol | X | | X | X | X | X | X | X | X | X | X |
| <b>Medication Review</b> | X | | X | X | X | X | X | X | X | X | X |
| <b>Quality of Life Assessments</b> | X | | | | - | X | | X | | | X |
| Subject Diary | $X^3$ | | | X | X | X | | X | | | X |
| Flexitouch Compliance | | | X | X | X | X | X | X | X | X | X |
| HCU, Adverse Events, & | | | X | X | X | X | X | X | X | X | X |
| <b>Device Observations</b> | | | | | | | | | | | |
| Flexitouch Training | | X | | | | | | | | | - |

<sup>&</sup>lt;sup>1</sup>Includes Lymphedema History

<sup>2</sup>Height and weight collected at Screening/Baseline, weight collected at all subsequent visits

<sup>3</sup>Dispense and train subject on subject diary completion

## 8.0 Study Device Accountability

To participate in the study, the Flexitouch must be covered by a payer. The Flexitouch will be provided to the subject and tracked according to normal business practices. Subjects' whose payer requires rental of the Flexitouch will be excluded from the study.

## 9.0 Risk Analysis and Adverse Events

#### 9.1 Risk Analysis

This study does not present risks above and beyond those normally associated with the use of this market cleared product. Pneumatic compression is a minimal risk therapy with minimal known complications or adverse events. However, as with any treatment, there is the possibility of undesirable events such as a local skin reaction to the device materials. The subject will be made aware of known complications at time of consent and monitored closely throughout the study.

Study subjects will be informed of any significant new findings that develop during the course of this study that may affect their willingness to continue participation. The principal investigator will oversee all safety aspects of the study and report all adverse events to the IRB per the IRB's reporting requirements. Should a subject choose to terminate his or her participation in the study, they will be treated according to the standard of care that applies at the point of withdrawal.

#### 9.2 Adverse Events

This study will collect device-related adverse events. A device related adverse event is defined as any untoward medical occurrence in a subject that is associated with the use of the Flexitouch device. If this device-related event is serious, investigators must report the event to Tactile Medical within 72 hours and to their IRB per their policy. A serious adverse event is defined as an event that, 1) results in death; 2) is life-threatening (places the subject at immediate risk of death from the experience as it occurred; 3) results in a persistent or significant disability/incapacity (substantial disruption of one's ability to carry out normal life functions); 4) results in medical or surgical intervention; 5) results in or prolongs existing hospitalization; 6) is medically unexpected, regardless of severity.

#### 10.0 Deviation from Study Plan

All deviations will be documented and reported to the IRB as required by IRB policies.

#### 11.0 Quality Assurance Procedures

This study will be conducted in accordance with Good Clinical Practice, Code of Federal Regulations (CFR), institutional research policies and procedures and other appropriate regulatory requirements to ensure subject safety and quality of clinical procedures related to the conduct of the clinical trial. As required by United States Food and Drug Administration (FDA) CFR (21 CFR 56) and the Declaration of Helsinki, the study protocol, amendments, and Informed Consent form will be reviewed and approved, according to 21 CFR §50 and §56, by each study center's IRB.

#### 11.1 Site Qualification

Tactile Medical personnel must conduct on-site Qualification Visits or a telephone qualification assessment to verify that there are adequate resources, staffing, and a sufficient subject pool to ensure successful enrollment and study completion.

#### 11.2 Data Collection Procedures

Raw data will be collected on appropriate source document worksheets, or site-specific appropriate forms which include but are not limited to, clinic charts and site-generated source document worksheets. If the site staff chooses to use site-specific data collection forms it may be beneficial for these to be reviewed by Tactile prior to use. Data collection shall be entered into the validated and secure Clindex electronic data capture systems.

#### 11.3 Clinical Site Monitoring

Clinical sites will be monitored for compliance with the clinical protocol, investigator agreement, and applicable regulations. Regular contact will be maintained to ensure:

- Subject safety
- That clinical site staff is well informed of regulations and sponsor requirements
- That the clinical protocol is followed
- That data is gathered in an accurate, complete and timely way
- That problems with data or data collection are addressed appropriately and in a timely manner
- That adverse events are properly reported in a timely manner

Investigator and Institution will permit trial related monitoring, audits, IRB review, and regulatory inspection(s), providing direct access to source data and documents as appropriate. Monitoring and source verification will be performed by Tactile Medical Clinical Research Associates (CRAs) and/or designee. Source verification includes reviewing subject source documentation and Case Report Forms (CRFs) for accuracy, completeness, and compliance with GCP procedures. In addition to site visits, a screening log must be submitted to Tactile Medical as requested (by fax or e-mail). This screening log should be reviewed with site staff to assess plan vs. actual recruitment.

### 11.4 Data Safety Monitoring

A periodic review may be completed by a designated member of the Scientific Advisory Board. The frequency of the review will be determined on a number of parameters including but not limited to: the rate of enrollment, number of complications, and number of significant deviations from the protocol. At the conclusion of the review the reviewer may provide recommendations that pertaining to study continuation, modification or termination of the trial, or a specific investigational site.

#### 11.5 Reports and Records

Records to be maintained by the investigator in a designated study file include:

- Investigational plan and all amendments
- Signed Investigator Agreement/Research Contract
- IRB approval letter, including a copy of the approved consent forms, progress reports, Adverse Event Report
- IRB roster or Assurance number, if applicable
- All correspondences relating to the conduct of this study between the site and sponsor, IRBs, and study monitor
- Curriculum Vitae and professional license for all study personnel, if applicable
- Site personnel signature and documentation regarding the Investigator's delegation of responsibility
- Clinical Site Visit log
- Protocol/device related training records for all applicable study personnel
- Screening log
- Reports (Table 4)

The following records must be maintained for each subject enrolled:

- Signed and dated informed consent forms
- Completed CRFs, queries, and source document worksheets (if applicable)
- Complete medical records including procedure reports, lab reports (as applicable), etc.

Investigators are required to prepare and submit to Tactile Medical or its designees complete, accurate, and timely reports on this investigation as required by regulations. The types of reports to be submitted are summarized in the table below.

Table 4: Investigator Reports

| Reports | Submit To | Timeframe |
|---|---|---|
| Serious Adverse Event | Sponsor and Reviewing | Sponsor: 72 hours |
| (SAE) | IRB | IRB: per their procedure |
| Withdrawal of IRB | Sponsor | Within 5 working |
| Approval | | Days |
| Progress | Sponsor and Reviewing IRB | Annually, at a |
| | | minimum |
| Final | Sponsor and | Within 3 months |
| | Reviewing IRB | following the |
| | | completion or termination of the |
| | | Investigator's part |

Subject study records, correspondence files, all supporting study documentation, and reports must remain on file at the investigational site for a minimum of ten years after the conclusion of this study. All investigators must contact Tactile Medical personnel prior to destroying or archiving off-site any records and reports pertaining to this study to ensure that they no longer need to be retained on-site. Additionally, Tactile Medical personnel must be contacted if the Investigator plans to leave the investigational site to ensure that arrangements for a new Investigator or records transfer are made prior to the Investigator's departure.

## 12.0 Change to Investigational Plan

Should changes in the study plan or protocol become necessary in the course of the clinical trial, proposed changes will be appropriately reviewed and approved by Tactile Medical personnel, Investigator, and appropriate IRB approval obtained before the any changes are implemented. All changes must be documented.

#### 13.0 Statistical Methods and Determination of Sample Size

#### 13.1 Statistical Analysis Plan

The analysis will be completed by a qualified statistician or analyst. The Sponsor will establish and maintain the trial database.

### 13.2 Determination of Sample Size

The study is planned to have up to 300 subjects enrolled. Each subject will undergo treatment as prescribed, using the Flexitouch system or Flexitouch Plus. This sample of convenience was selected based on the investigator's previous pilot study and experience with this patient population.

#### 14.0 Compensation

Study subjects may be compensated for their time and travel for participating in this study.

#### 15.0 Publication Plan

All information obtained during the conduct of the study will be considered to be confidential and is the property of Tactile Medical. Written permission from Tactile Medical personnel must be obtained before disclosing any information related to this study. All publications (e.g. manuscripts, abstracts, and slide presentations) based on this study must be submitted to Tactile Medical for review and approval before submission or according to the individual site clinical trial agreement.

#### 16.0 References

- 1. Jensen MR, Simonsen L, Karlsmark T, Bulow J. Lymphoedema of the lower extremities--background, pathophysiology and diagnostic considerations. Clin Physiol Funct Imaging. 2010 Nov;30(6):389-98.
- 2. Cormier JN, Askew RL, Mungovan KS, Xing Y, Ross MI, Armer JM. Lymphedema beyond breast cancer: a systematic review and meta-analysis of cancer-related secondary lymphedema. Cancer. 2010 Nov 15:116(22):5138-49.
- 3. Todo Y, Yamamoto R, Minobe S, Suzuki Y, Takeshi U, Nakatani M, et al. Risk factors for postoperative lower-extremity lymphedema in endometrial cancer survivors who had treatment including lymphadenectomy. Gynecol Oncol. 2010 Oct;119(1):60-4.

- 4. Langbecker D, Hayes SC, Newman B, Janda M. Treatment for upper-limb and lower-limb lymphedema by professionals specializing in lymphedema care. Eur J Cancer Care (Engl). 2008 Nov;17(6):557-64.
- 5. Mayrovitz HN. Interface pressures produced by two different types of lymphedema therapy devices. Phys Ther. 2007 Oct;87(10):1379-88.
- 6. Ridner SH, McMahon E, Dietrich MS, Hoy S. Home-based lymphedema treatment in patients with cancer-related lymphedema or noncancer-related lymphedema. Oncol Nurs Forum. 2008 Jul;35(4):671-80.
- 7. Wilburn O, Wilburn P, Rockson SG. A pilot, prospective evaluation of a novel alternative for maintenance therapy of breast cancer-associated lymphedema [ISRCTN76522412]. BMC Cancer. 2006;6:84.
- 8. Cannon S. Pneumatic compression devices for in-home management of lymphedema: two case reports. Cases J. 2009;2:6625.
- 9. Keeley V, Crooks S, Locke J et al. A quality of life measure for limb lymphoedema (LYMQOL), J Lymphedema, 2010, 5(1)

## 17.0 Appendices

Appendix A: Lymphedema Quality of Life Tool (LYMQOL)

Appendix B: SF-36 Health Survey v.2 (SF-36)

Appendix C: Subject Diary

# Appendix A: Lymphedema Quality of Life Tool (LYMQOL)

| LYMQOL (Source Document) Assessment of Quality of Life Changes on Lower Extremity Lymphe Pneumatic Compression Device at Home Protocol #5010 | edema Pati | ents using a | an Advance | d |
|---|---|---|---|---|
| Subject ID: Visit Date:/ | | | | |
| <u>LYMQOL LEG</u><br>Lymphoedema Quality of Life Tool | | | | |
| This questionnaire has been designed and validated for patie lymphoedema of one or both legs to measure quality of life. Please tick the box that best describes how you feel about ea | | | | |
| If any of the items are not applicable to you, please write N/A in the relevant answer box(es) | | | | |
| (Q1) How much does your swollen leg affect the following activities? | Not at all | A little | Quite a bit | A lot |
| a) your walking | | | | |
| b) your ability to bend, e.g. to tie shoelaces or cut toenails | | | | |
| c) your ability to stand. | | | | |
| d) your ability to get up from a chair. | | | | |
| e) your occupation | | | | |
| f) your ability to do housework | | | | |
| | Not at | A little | Quite a | A lot |
| (Q2)Does the swelling affect your leisure activities/<br>social life? | 33,6 34/37 | | State County | |
| Please give examples of this | | | | |
| | Not at all | A little | Quite a bit | A lot |
| (Q3) How much do you have to depend on other people? | | | | |
| (Q4) How much do you feel the swelling affects your appearance? | | | | |
| (Q5) How much difficulty do you have finding clothes to fit? | | | | |
| (Q6) How much difficulty do you have finding clothes you would like to wear? | | | | |
| (Q7) Do you have difficulty finding shoes to fit? | | | | |
| (Q8) Do you have difficulty finding socks/ tights/<br>stockings to fit? | | | | |
| (Q9) Does the swelling affect how you feel about yourself? | | | | |

(Q11) Does your lymphoedema cause you pain?

(Q10)Does it affect your relationships with other people?

| Assessment of Quality of Life Changes on Lower Extremity L<br>Advanced Pneumatic Compression Device at Home | .ympheder | na Patient | s using an | |
|---|---|---|---|---|
| Protocol #5010 | | | | |
| Subject ID: | | | | |
| | Not at | A little | Quite a | A lot |
| | all | | bit | |
| Q12) Do you have any numbness in your swollen leg(s)? | | | | |
| Q13) Do you have any feelings of "pins & needles" or ingling in your swollen leg(s) | | | | |
| Q14) Does (do) your swollen leg(s) feel weak? | | | | |
| Q15) Does (do) your swollen leg(s) feel heavy? | | | | |
| 4 | NI-4-4 | A 1:44 | 0 | LA 1-4 |
| the past week | Not at | A little | Quite a<br>bit | A lot |
| Q16) Have you had trouble sleeping? | | | | |
| Q17) Have you had difficulty concentrating on things,<br>g. reading? | | | | |
| 218) Have you felt tense? | | | | |
| 219) Have you felt worried? | | | | |
| Q20) Have you felt irritable? | | | | |
| Q21) Have you felt depressed? | | | | |
| Q22) Overall, how would you rate your quality of life at pro<br>Please mark your score on the following scale: | esent? | | | |
| | 8=8 88 | 9 | 10 | |
| 0 1 2 3 4 5 6<br>poor | 7 8 | 3 | excellent | |
| poor Thank you for completing this If you have any comments or queries about it, please discuss | form.<br>these wit | h your stu | ıdy coordin | ator |
| poor Thank you for completing this | form.<br>these wit<br>nission fro | h your stu | ıdy coordin | ator |
| Thank you for completing this If you have any comments or queries about it, please discuss Questions 16 to 21 have been reproduced with perm | form. these wit nission fro 30 Quest y provided t | h your stum the EC ionnaire. hat this copichanges are be forwarde | ordin<br>PRTC.<br>yright statem<br>e made withoud in writing to | ent is<br>ut<br>o Dr |
| Thank you for completing this of you have any comments or queries about it, please discuss Questions 16 to 21 have been reproduced with permoduced with permoduced with permoduced with permoduced freely a part of the QLQ-C Copyright November 2007 Ref. LEG V II All rights reserved. This document can be used or reproduced freely left intact, that the source is acknowledged, that the user registers a permission of the author. Application for permission and for registrativaughan Keeley, Consultant in Palliative Medicine, Nightingale Mac | form. these wit nission fro 30 Quest y provided t and that no tion should emillan Unit | h your stum the EC ionnaire. hat this copchanges are be forwarded, 117A Lond | ordin<br>PRTC.<br>yright statem<br>e made withoud in writing to | ent is<br>ut<br>o Dr<br>rby |

Version 2.0 November 2007 (Format updated 16Oct2018)


## Appendix B: SF-36 Health Survey v.2 (SF-36)

| Assessm | tic Compression D | ife Changes on i | Lower Extremity Lyr | mphedema Patieni | ts using an Advan | ced |
|---|---|---|---|---|---|---|
| Subje | ect ID: | | Ir | nitial Report Dat | e://<br>(ddMMMyyyy) | |
| Study \((select on | | eline Visit | ☐ Week 12 Vi | sit | ☐ Week 24 Vi | sit |
| | You | r Hea | lth and | Well-F | Being | |
| keep ti | | ou feel and h | about your hea<br>now well you and<br>arvey! | | | 100 |
| | ch of the follo | | ons, please mai | rk an 🔀 in th | e one box tha | t best |
| 1. In | general, woul | d you say yo | our health is: | | | |
| | Excellent | Very good | Good | Fair | Poor | |
| | | <b>▼</b> □ 2 | <b>▼</b> 3 | 4 | <b>▼</b> 5 | |
| 2. <u>Co</u> | | <u>e vear ago,</u> l | 10w would you | rate your hea | alth in genera | 1 |
| | Much better<br>now than one<br>year ago | Somewhat<br>better<br>now than one<br>year ago | About the same as one year ago | Somewhat<br>worse<br>now than one<br>year ago | Much worse<br>now than one<br>year ago | |
| | <b>▼</b> | <b>▼</b> □ 2 | <b>▼</b> 3 | <b>▼</b> □ 4 | <b>▼</b> | |

| Ass<br>Pne | -36v2 (Source Document)<br>essment of Quality of Life Changes on Lower Extremity Lymph<br>umatic Compression Device at Home<br>locol #5010 | edema Patieni | ts using an Ad | vanced |
|---|---|---|---|---|
| S | ubject ID: | | | |
| 3. | The following questions are about activities ye day. Does your health now limit you in these | | | |
| | | Yes,<br>limited<br>a lot | Yes, limited a little | No, not limited at all |
| a | <u>Vigorous activities</u> , such as running, lifting heavy objects, participating in strenuous sports | 1 | 2 | 3 |
| b | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 1 | 2 | 3 |
| c | Lifting or carrying groceries | I | 2 | 3 |
| d | Climbing several flights of stairs | 1 | 2 | 3 |
| е | Climbing one flight of stairs | 1 | 2 | |
| f | Bending, kneeling, or stooping | i | 2 | |
| g | Walking more than a mile | ī | 2 | 3 |
| h | Walking several hundred yards | 1 | 2 | |

| Asse<br>Pne | -36v2 (Source Documen<br>essment of Quality of Life Changes<br>umatic Compression Device at Ho.<br>ocol #5010 | on Lower Extr | emity Lymphe | dema Patients | using an Adva | nced |
|---|---|---|---|---|---|---|
| S | Subject ID: | | | | | |
| 4. | During the past 4 weeks, following problems with result of your physical he | your work | | | | |
| | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| а | Cut down on the <u>amount of time</u> you spent on work or other activities | 1 | 2 | 3 | 4 | 5 |
| Ъ | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| c | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 4 | 5 |
| d | Had <u>difficulty</u> performing the work or other activities (for example, it took extra effort) | 1 | 2 | 3 | 4 | 5 |
| 5. | During the <u>past 4 weeks</u> , following problems with <u>result of any emotional p</u> | your work | or other re | gular daily | activities <u>a</u> | is a |
| | | All of the time | | Some of the time | A little of the time | None of the time |
| a | Cut down on the <u>amount of time</u> you spent on work or other activities | 1 | 2 | 3 | 4 | 5 |
| b | Accomplished less than you would like | i | 2 | 3 | 4 | 5 |
| ¢ | Did work or other activities less carefully than usual | i | 2 | 3 | 4 | 5 |

| SI -30 VZ (Oddice Document | SF-36v2 | (Source | Document |
|----------------------------|---------|---------|----------|
|----------------------------|---------|---------|----------|

Assessment of Quality of Life Changes on Lower Extremity Lymphedema Patients using an Advanced Pneumatic Compression Device at Home Protocol #5010

Subject ID: \_\_\_\_ - \_\_\_ -

6. During the <u>past 4 weeks</u>, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups?

| Not at all | Slightly | Moderately | Quite a bit | Extremely |
|------------|----------|------------|-------------|-----------|
| • | | lacksquare | | • |
| <u> </u> | 2 | 3 | 4 | 5 |

7. How much bodily pain have you had during the past 4 weeks?

| None | Very mild | Mild | Moderate | Severe | Very severe |
|------|------------|------|----------|----------|-------------|
| | lacksquare | | | | |
| i i | 2 | | <u> </u> | <u> </u> | 6 |

8. During the <u>past 4 weeks</u>, how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)?

| Not at all | A little bit | Moderately | Quite a bit | Extremely |
|------------|--------------|------------|-------------|-----------|
| ▼<br>□ 1 | ▼<br>□ 2 | <b>▼</b> | <b>▼</b> | <b>▼</b> |

| Asses<br>Pneui | <b>36v2</b> (Source Document) ssment of Quality of Life Changes of matic Compression Device at Homocol #5010 | on Lower Extre | emity Lymphed | lema Patients | using an Advar | nced |
|---|---|---|---|---|---|---|
| Su | ıbject ID: | <del>-</del> | | | | |
| 9 | These questions are about during the past 4 weeks. I comes closest to the way y during the past 4 weeks | For each qu | iestion, ple | ase give tl | he one answ | er that |
| | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| a | Did you feel full of life? | ī | 2 | 3 | 4 | 5 |
| ъ | Have you been very nervous? | Т | 2 | 3 | 4 | 5 |
| 3 | Have you felt so down in the dumps that nothing could cheer you up? | 1 | 2 | 3 | 4 | 5 |
| | Have you felt calm and peaceful? | 1 | 2 | 3 | 4 | 5 |
| е | Did you have a lot of energy? | 1 | 2 | 3 | 4 | 5 |
| f | Have you felt downhearted and depressed? | 1 | 2 | 3 | 4 | 5 |
| g | Did you feel worn out? | 1 | 2 | 3 | 4 | 5 |
| h | Have you been happy? | 1 | 2 | 3 | 4 | 5 |
| í | Did you feel tired? | ī | 2 | 3 | 4 | 5 |
| 9 | During the <u>past 4 weeks,</u> h<br>emotional problems intert<br>friends, relatives, etc.)? | | | | | |
| | All of Most of the time the time | | | little of ne time | None of the time | |

Version: A 18Dec2014 (Format updated 16Oct18)

Confidential Source

1 2 3


4 5

| SF-36v2 (Source Documen<br>Assessment of Quality of Life Changes<br>Pneumatic Compression Device at Hol<br>Protocol #5010 | on Lower Extre | emity Lymphe | dema Patients | s using an Adv | /anced |
|---|---|---|---|---|---|
| Subject ID: | <del></del> | | | | |
| 11. How TRUE or FALSE is | each of the | following | statement | s for you? | |
| | Definitely true | Mostly true | Don't<br>know | Mostly false | Definitely false |
| I seem to get sick a little easier than other people | 1 | 2 | 3 | 4 | 5 |
| ь I am as healthy as<br>anybody I know | 🔲 т | 2 | 3 | 4 | 5 |
| I expect my health to get worse | 🔲 т | 2 | 3 | 4 | 5 |
| d My health is excellent | 1 i | 2 | 3 | 4 | 5 |
| Signature of person completing: | | | Dat | te:/_ | |
| | | | | Day Mo | onth Year |

Thank you for completing these questions!

Version: A 18Dec2014 (Format updated 16Oct18)

Confidential Source


## **Appendix C: Subject Diary**

| SUBJECT DIA | ARY | Prescription | on: | | | | |
|---|---|---|---|---|---|---|---|
| Subject ID: | | Flexitouch_ | | Actitouch | Comp | ression Stockin | gs |
| | | MC | NTH: | | | | |
| | Sunday | Monday | Tuesday | Wednesday | Thursday | Friday | Saturday |
| Check<br>treatments<br>used each<br>day | □ None □ Flexitouch □ Actitouch □ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings |
| Check<br>treatments<br>used each<br>day | □ None □ Flexitouch □ Actitouch □ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings |
| Check<br>treatments<br>used each<br>day | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings |
| Check<br>treatments<br>used each<br>day | □ None □ Flexitouch □ Actitouch □ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | ☐ None ☐ Flexitouch ☐ Actitouch ☐ Compression Stockings |
| Check<br>treatments<br>used each<br>day | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings | □ None □ Flexitouch □ Actitouch □ Compression Stockings |
| SUBJECT SIG | SNATURE: | | | | DATE:_ | | |
| Reminder: ` | Your next ap | pointment is | scheduled 1 | for: | | Version | 3.1, July 2019 |